CLINICAL TRIAL: NCT04492267
Title: SARS-CoV-2 Infection in Patients From Two Tertiary Inflammatory Bowel Disease (IBD) Centres: Frequency of Suspected and Confirmed Infections, Severity and Outcome Management
Brief Title: Inflammatory Bowel Disease (IBD) and Covid-19 Infection
Acronym: MICI-Covid-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7930
Record Dates: First submitted 2020-07-23; First posted 2020-07-30 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Inflammatory Bowel Disease
Keywords: SARS-CoV-2; Inflammatory Bowel Disease; IBD; Crohn's disease; Ulcerative colitis; Immunosuppressant therapy; Biologicals; Severe respiratory disease; intensive care unit; Mechanical ventilation; Death
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative; Respiration Disorders; Death

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Most of the inflammatory bowel disease (IBD: Crohn's disease and ulcerative colitis) in a tertiary expert Centre are on immunosuppressive and/or biological therapy. Theoretically, these treatments may increase patients' risk of infection, in particular viral infection. Therefore, the current SARS-Cov-2 pandemia, with its unprecedent worldwide morbidity and mortality, may have a negative impact on IBD patients' clinical course. Identifying an increased risk in this particular patients' population as well as the risk/protective factors is of outstanding importance, in order to adapt their treatment and surveillance. As a consequence, our aims were (i) to measure retrospectively the risk of SARS-CoV-2 (proven by biological testing or suspected due to record of potential clinical symptoms of COVID-19 infection) in this patients' cohort (principal objective), (ii) to identify risk or protective factors for SARS-CoV-2 infection in IBD, and (iii) to analyze the outcome of patients in case of suspected or confirmed COVID-19. The results of this study may be important to adjust our surveillance and therapeutic strategy in these patients, in particular if high virus circulation will occur in the future.

ELIGIBILITY:
Inclusion Criteria:

* Patient over the age of 18 years
* IBD patients (Crohn's disease, ulcerative colitis, indeterminate colitis)
* Patient agreeing to participate in the study

Exclusion Criteria:

* Patient unable to understand the study protocol or to answer simple anamnestic questions due to language barrier
* Patient under guardianship or trusteeship
* Patient under safeguard of justice

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: IBD patient (Crohn's disease, ulcerative colitis, indeterminate colitis) over the age of 18 years
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2020-07-07 (Actual); Primary Completion 2021-01-07 (Estimated); Study Completion 2021-01-07 (Estimated)

PRIMARY OUTCOMES:
Retrospective analysis of severity and specific needs in case of SARS-CoV-2 infection in IBD patients | Files analysed retrospectily from March 1st, 2020 to July 31, 2020 will be examined

CONTACTS AND LOCATIONS:
Locations (1):
- Service Hépato-Gastroentérologie et Assistance Nutritive Hôpitaux Univesitaires de Strasbourg, Strasbourg, France